CLINICAL TRIAL: NCT00975416
Title: Oxytocin and Cognitive Behavioral Therapy in Drug Dependence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999908432; 08-DA-N432
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Drug Dependence
Keywords: Drug Dependence; Cognitive Behavior; Oxytocin; Cocaine; Heroin; fMRI
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

ARMS (3):
- Methadone (Placebo Comparator): Intranasal oxytocin administered in the context of cognitive behavioral therapy to methadone dependent outpatients
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Intranasal Oxytocin; Drug: Placebo
- Outpatient Cocaine (Placebo Comparator): Intranasal oxytocin administered in the context of cognitive behavioral therapy to cocaine dependent outpatients
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Intranasal Oxytocin; Drug: Placebo
- Inpatient Cocaine (Placebo Comparator): Intranasal oxytocin administered in the context of cognitive behavioral therapy to cocaine dependent inpatients
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Intranasal Oxytocin; Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Intranasal oxytocin given in the context of cognitive behavioral therapy
Drug: Intranasal Oxytocin — Intranasal oxytocin given in the context of cognitive behavioral therapy
Drug: Placebo — Placebo given in the context of cognitive behavioral therapy

SUMMARY:
Background:

- The therapeutic alliance between therapist and patient may contribute to favorable outcomes in all types of psychotherapy, including cognitive behavioral therapy (CBT) for drug dependence. Oxytocin, a hormone and neurotransmitter, has been shown to increase trust in other people and may reduce stress and improve comfort in social situations by decreasing the sensation of social anxiety. Researchers are interested in determining if oxytocin can improve the outcomes of therapy for drug dependence by strengthening perceived levels of trust between therapist and patient.

Objectives:

- To determine whether oxytocin enhances the therapeutic alliance and treatment retention for CBT for drug use.

Eligibility:

- Individuals between 18 and 65 years of age who are healthy volunteers with no history of drug abuse, participants in outpatient or inpatient treatment programs for cocaine use, methadone-dependent participants in a treatment program, or non-treatment-seeking cocaine users.

Design:

* Participants in each treatment arm who comply with the study requirements will be randomly assigned to receive one dose of oxytocin or placebo approximately 1 hour before each weekly CBT session.
* The outpatient treatment intervention will be 12 weeks of weekly individual CBT. The inpatient treatment intervention will be 6 weeks of twice-weekly individual CBT sessions. Sessions will be audiotaped. Participants and counselors will be told that the sessions are to be taped.
* During treatment, participants will provide urine and breath samples under staff observation. Participants will also complete questionnaires about mood and mental health, provide other samples as required, and participate in computerized psychological testing as directed by researchers.

DETAILED DESCRIPTION:
Objective The therapeutic alliance (TA), a working relationship between therapist and patient, may contribute to favorable outcomes in all types of psychotherapy, including cognitive-behavioral therapy (CBT) for drug dependence. Enhancement of the TA may be possible through intranasal administration of the hormone and neurotransmitter oxytocin, which is associated with social bonding and trust. The objective of this study is to determine whether addition of intranasal oxytocin to a course of CBT for drug dependence enhances TA and treatment retention and reduces drug use post-treatment. The study will assess changes in performance on tasks that probe decision-making, emotional processing, and drug-cue reactivity. We will employ fMRI on a subset of participants to study the neural correlates of these processes.

Study population. The treatment portion of the study will be conducted in three parallel arms, not intended to be statistically compared to each other: (1) Outpatient Methadone arm (physically dependent heroin users, n = 80 evaluable); (2) Outpatient Cocaine arm (cocaine-dependent individuals, non-opiate-dependent, n = 80 evaluable); 3) Inpatient Cocaine arm (cocaine-dependent individuals, non-opiate-dependent, n = 80 evaluable). There will also be two groups of non-treatment-seeking controls (20 cocaine-using, 20 non-drug-using) to rule out practice effects on tasks; controls will not receive oxytocin or CBT.

Experimental design and methods. Primary outcome measures will be TA in all arms and drug use for methadone and cocaine outpatient arms. (1) Methadone arm: after a 5-week baseline for stabilization on methadone, participants will undergo 12 weeks of CBT, with random assignment to oxytocin (24 IU, administered before each session) or placebo. (2 and 3) Cocaine arms, inpatient and outpatient: after a 1-week baseline for assessment of drug use, participants will undergo 6 and 12 weeks respectively of CBT, with random assignment to oxytocin (24 IU, administered before each session) or placebo.

Outcome measures: Principle outcome measures for the outpatient arms will be TA measured at several points during CBT, treatment retention, and attendance at CBT sessions. Secondary outcome measures are drug use during treatment and at follow-up, drug craving during treatment and at follow-up, stress reduction during treatment and at follow-up, HIV risk behaviors during treatment and at follow-up, behavioral performance on various tasks, and neural response to these tasks for the imaging subgroup. The outcome measures for the inpatient arm will be the same as for the outpatient arms with the exception of drug use during treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must:

1. Be between age 18 and 65.
2. Methadone arm only: opiate dependence for the past year determined by clinical exam, opiate-positive urine during screening and diagnosis confirmed by SCID.
3. Cocaine outpatient arm: cocaine dependence determined by clinical exam, cocaine-positive urine during screening and diagnosis confirmed by SCID.
4. Cocaine inpatient arm: Cocaine dependence determined by clinical exam during screening and diagnosis confirmed by SCID.
5. Control participants: cocaine dependent and non-drug using, will be recruited to provide appropriate matches for subjects in the two treatment arms with respect to the following characteristics: age, gender, IQ, socioeconomic factors, and years of education.
6. Be free of dependence on other substances except nicotine, heroin (for the methadone arm only), or cocaine at the time of participation. Justification: Dependence on other substance may result in unique CNS deficits that would confound our results. Nicotine dependence will be allowed because nicotine use is not associated with a drug high in normal usage and the prevalence of nicotine dependence in cocaine users may make it impractical to exclude nicotine users. While it might be preferable to exclude individuals whose use of other substances reaches the threshold of abuse, inclusion of such individuals will not necessarily contaminate the data. Inpatient cocaine arm subjects who meet DSM-IV TR criteria for the course specifier In a Controlled Environment may have a history of dependence on substances other than cocaine before their admission to the inpatient treatment program. Assessment tool(s): SCID with confirmation by negative urine drug screen.

   For participation in the scanning portion of the study, participants must also:
7. Be between the ages of 18-55. Justification: Many of the cognitive processes under study change with age. In addition, the risk of difficult-to-detect medical abnormalities such as silent cerebral infarcts increases with age. Individuals over 55 will therefore be excluded. Assessment tool(s): driver s license, birth certificate, or other government-issued form of identification.
8. Be in good health. Justification: Many illnesses can alter fMRI signal and alter cognition. Assessment tool(s): Participants will provide a brief health history during phone screening, and undergo a history and physical examination with a qualified IRP clinician (exam details discussed below in reference to specific exclusion criteria).
9. Be right-handed. Justification: Many of the brain functions to be assessed in this protocol have shown some evidence of being lateralized in the brain. In order to reduce variability in the data, participants must be right-handed. Assessment tool(s): Edinburgh Handedness Inventory.

EXCLUSION CRITERIA:

Participants will be excluded if they have evidence of:

1. Schizophrenia or any other DSM-IV psychotic disorder; history of bipolar disorder; current major depressive disorder.
2. Current dependence on alcohol or sedative-hypnotic, e.g. benzodiazepine (by DSM-IV criteria), except for inpatient cocaine arm.
3. Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires.
4. Renal insufficiency with serum creatinine greater than 1.7.
5. Medical illness that in the view of the investigators would compromise participation in research such as: a history of syncope, family history of sudden death, electrolyte imbalance, bradycardia, arrhythmias, marked sustained high BP with SBP > 160 and or DBP > 100 on more than two readings without 3rd reading being below these parameters and not stabilized on antihypertension medications before the starting the study, congestive heart failure, history or finding on screening EKG of significant abnormality such as prolonged QTc (> 450ms) , or AIDS or HIV positive with T cell count less than or equal to 200.
6. Urologic conditions that would inhibit urine collection.
7. Untreated Endocrine disorders.
8. Pregnancy, planning to become pregnant, or breastfeeding. In addition, women of child-bearing age who are sexually active are required to use an effective form of birth control for the duration of the study. Effective forms of birth control include:

   1. hormonal contraceptives (birth control pills, injectable hormones, vaginal ring hormones),
   2. surgical sterility (tubal ligation or hysterectomy)
   3. IUD
   4. Diaphragm with spermicide
   5. Condom with spermicide
9. For the methadone arm, use of any drugs that would interact with methadone to produce adverse effects such as Class I or Class III antiarrhythmics, TCA s, MAOI s, calcium channel blockers, neuroleptics or frequent use of sedative hypnotic drugs. Justification: Avoidance of adverse interaction with methadone. Assessment tool(s): Clinical interview and tox screen.
10. Use of any drugs (prostaglandins, vasoconstricting agents or anesthetic medications, for example) that may interact with oxytocin. Justification: Avoidance of adverse interaction with oxytocin. Assessment tool(s): Clinical interview and tox screen
11. History of hypersensitivity to oxytocin or vehicle, i.e. propylparahydroxybenzioate, methylparahydroxybenziate, chlorbutanol hemihydrate. Assessment tool: clinical interview
12. Presence of or history of clinically significant allergic rhinitis as assessed by MRP or PI. Justification: Inflammation of nasal mucosa could interfere with mucosal absorption of intranasally administered OT.

    In addition, participants will be excluded from fMRI scanning if they:
13. Are not suitable for fMRI due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia. Justification: MR scanning is the primary measurement tool used in this portion of the protocol. Assessment tool(s): Prospective participants will fill out an MRI screening questionnaire and undergo an interview with an MR technologist. Pregnancy tests will be performed on all female participants of childbearing age before each experimental session. Questions concerning suitability for scanning will be referred to the MR Medical Safety Officer. Prospective participants will be questioned about symptoms of claustrophobia and placed in the mock scanner during their screening visit to assess for possible difficulty tolerating the confinement of the scanner and for ability to physically fit into the scanner.
14. Have coagulopathies, history of or current superficial or deep vein thrombosis, or musculoskeletal abnormalities restricting ability to lie flat for extended periods. Justification: MR scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately two hours. Therefore, conditions that would make that difficult (e.g. chronic back pain, significant scoliosis) or dangerous (e.g. familial hypercoagulability syndrome, history of thrombosis) will be exclusionary. Assessment tool(s): History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to assess comfort issues.
15. Have HIV or syphilis. Justification: HIV and syphilis can both have CNS sequelae, thus introducing unnecessary variability into the data. Assessment tool(s): HIV blood test, syphilis serology (positive FTA).
16. Have any neurological illnesses. This includes, but is not limited to, seizure disorders, migraine, multiple sclerosis, movement disorders, or history of head trauma, CVA, or CNS tumor. Justification: CNS diseases alter CNS function and, possibly, the neuronal-vascular coupling that forms the basis of the BOLD fMRI signal to be used in this study. Assessment tool(s): History and physical examination by a qualified IRP clinician, urine drug screening for anticonvulsants not disclosed by history. History of head trauma with loss of consciousness of more than 5 minutes or with postconcussive sequelae lasting more than two days, regardless of loss of consciousness, will be exclusionary.
17. Regularly use any prescription, over-the-counter, or herbal medication that may alter CNS function, cardiovascular function, or neuronal-vascular coupling. Justification: Compounds that alter BOLD signal will alter the primary measure used in the study. Assessment tool(s): History and comprehensive urine drug screening to detect use of antidepressants, benzodiazepines, antipsychotics, anticonvulsants, barbiturates, and other common medications and drugs of abuse.

All participants who are fullfill criteria for fMRI scanning will be asked to undergo scanning; we anticipate that approximately 50 percent of enrolled participants will be scanned.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Lee, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Aharon I, Etcoff N, Ariely D, Chabris CF, O'Connor E, Breiter HC. Beautiful faces have variable reward value: fMRI and behavioral evidence. Neuron. 2001 Nov 8;32(3):537-51. doi: 10.1016/s0896-6273(01)00491-3. PMID 11709163
- [Background] Amico JA, Mantella RC, Vollmer RR, Li X. Anxiety and stress responses in female oxytocin deficient mice. J Neuroendocrinol. 2004 Apr;16(4):319-24. doi: 10.1111/j.0953-8194.2004.01161.x. PMID 15089969
- [Background] Anderson-Hunt M, Dennerstein L. Increased female sexual response after oxytocin. BMJ. 1994 Oct 8;309(6959):929. doi: 10.1136/bmj.309.6959.929. No abstract available. PMID 7950665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at an inpatient treatment center. Screening was included in the study. Also, baseline characterization was done as a within subject study with tasks and measures before randomization to oxytocin or placebo and treatment with cognitive behavioral therapy.
  Methadone and outpatient cocaine arms did not recruit participants.
Pre-assignment Details: 63 participants were screened, 30 were randomized. Subjects completed a battery of tasks and measures on oxytocin and on placebo before entering into randomized treatment phase where they were assisgned to the oxytocin or placebo arm with all subjects receiving cognitive behavioral therapy during the treatment phase.
Groups:
- Inpatient Cocaine Oxytocin: Intranasal oxytocin administered in the context of cognitive behavioral therapy to cocaine dependent inpatients
  Oxytocin Nasal Spray: Intranasal oxytocin given in the context of cognitive behavioral therapy
- Inpatient Cocaine Placebo: Placebo administered in the context of cognitive behavioral therapy to cocaine dependent inpatients Placebo given in the context of cognitive behavioral therapy
Period: Overall Study
Arm/Group | Inpatient Cocaine Oxytocin | Inpatient Cocaine Placebo
Started | 14 | 16
Completed | 11 | 11
Not Completed | 3 | 5
Not completed — early discharge from tx | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Inpatient Cocaine Placebo: Intranasal placebo administered in the context of cognitive behavioral therapy to cocaine dependent inpatients
  Intranasal Placebo given in the context of cognitive behavioral therapy
- Total: Total of all reporting groups
Arm/Group | Inpatient Cocaine Oxytocin | Inpatient Cocaine Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.2) | 40.8 (10.0) | 40.9 (9.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Alliance
Description: Penn Helping Alliance Questionnaire containing 19 questions with possible scores from 19(low therapeutic alliance)-114(high therapeutic alliance).
  Working Alliance Inventory containing 36 questions with possible scores from 36(low therapeutic alliance)-252 (high therapeutic alliance).
Time Frame: Post 12 weeks treatment with cognitive behavioral therapy
Population: Number of participants for analysis was determined by the number of participants who had post-treatment outcome measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inpatient Cocaine Oxytocin | Inpatient Cocaine Placebo
Number analyzed (Participants) | 14 | 16
units on a scale
  Working Alliance Inventory | 220.43 (20.55) | 223.13 (41.81)
  Penn Helping Alliance Questionnaire | 99.23 (8.45) | 99.81 (10.12)
Statistical Analysis 1: Comparison: Inpatient Cocaine Oxytocin vs Inpatient Cocaine Placebo; Repeated measures ANOVA to deterimine whether oxytocin increased compared to placebo measures of therapeutic alliance (as measured by the Helping alliance questionnaire) pre compared to post 12 sessions of CBT; Test type: Superiority or Other; p = 0.927, ANOVA
Statistical Analysis 2: Comparison: Inpatient Cocaine Oxytocin vs Inpatient Cocaine Placebo; Repeated measures anova to determine if oxytocin compared to placebo increased therpeutic alliance as measured by the working alliance inventory after 12 sessions of CBT; Test type: Superiority or Other; p = 0.60, ANOVA

2. Other Pre Specified Outcome: Drug Craving
Description: Cocaine Craving Questionnaire
Time Frame: Post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Methadone: Intranasal oxytocin administered in the context of cognitive behavioral therapy to methadone dependent outpatients
  Oxytocin Nasal Spray: Intranasal oxytocin given in the context of cognitive behavioral therapy
- Outpatient Cocaine: Intranasal oxytocin administered in the context of cognitive behavioral therapy to cocaine dependent outpatients
  Oxytocin Nasal Spray: Intranasal oxytocin given in the context of cognitive behavioral therapy
- Inpatient Cocaine: Intranasal oxytocin administered in the context of cognitive behavioral therapy to cocaine dependent inpatients
  Oxytocin Nasal Spray: Intranasal oxytocin given in the context of cognitive behavioral therapy
Arm/Group | Methadone | Outpatient Cocaine | Inpatient Cocaine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/28
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/28

LIMITATIONS AND CAVEATS:
1 participant committed suicide outside of that occurred outside of adverse event time frame.

There were 12 occurrences of computer malfunction during the study. This did not effect data collection for primary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No